CLINICAL TRIAL: NCT02912039
Title: Electromyographic Assessment of the TetraGraph in Normal Volunteers
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, J. Ross Renew, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 16-005022
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2023-05-17 (Actual); Status verified 2018-07

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: TetraGraph — A sequence of 3 sets of Train of four (TOF) stimuli delivered (every 20 sec) at the pre-determined current amplitude (for instance, 40 mA, then 30 mA, then 50 mA, then 20 mA).
Device: TOF Watch — A sequence of 3 sets of TOF stimuli delivered (every 20 sec) at the pre-determined current amplitude (for instance, 40 mA, then 30 mA, then 50 mA, then 20 mA).

SUMMARY:
There is an urgent need for an easy-to-use and accurate quantitative neuromuscular monitor in the clinical setting. The aim of this clinical investigation is to examine a prototype of a quantitative monitoring instrument that will meet most, if not all, of the clinical requirements.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 years or older
2. Volunteer meets the American Society of Anesthesiology (ASA) physical status I-III criteria
3. Volunteer has provided verbal informed consent

Exclusion Criteria

1. Presence of an underlying neuromuscular disease
2. Use of medications known to interfere with neuromuscular transmission
3. Volunteer has open sores/rashes at the locations needed for electrode application
4. Volunteer does not tolerate a trial electrical stimulation comfortably.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population for this study is normal, healthy, unpremedicated human volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Comparison of train of four measurements between TOF Watch and TetraGraph | During stimulation
  The primary endpoint will be an analysis of the agreement between the TOF-Watch (the current gold standard) and TetraGraphTM devices during neuromuscular monitoring. Data Acceleromyography (AMG) and Electromyography (EMG) will be compared between the two devices during testing of single twitch (ST) and train of four (TOF) patterns at varying current amplitudes, from threshold amplitude (the lowest current amplitude that is able to generate a muscle response), to supramaximal current amplitude (the amplitude that elicits maximal muscle response). Bias and limits of agreement will be calculated for each stimulation pattern (ST and TOF) at currents between submaximal and supramaximal amplitude. Measured responses obtained with the two technologies (AMG and EMG) will be compared.

SECONDARY OUTCOMES:
Noise level | During stimulation
  Acceptable levels of electrical noise when no stimulus is being applied (random noise, power-line noise, and background EMG recorded in a relaxed volunteer with low recording electrode impedance should be 0.2 mV RMS or less).
Stimulus artifact | During stimulation
  That the stimulus artifact will not obscure the EMG response when a stimulus is applied.
Appearance EMG response | During stimulation
  Appearance of an EMG response at threshold stimulation levels, enough to just barely elicit a visible twitch response and elicit measurable acceleration on the TOF-Watch.
EMG amplitude | During stimulation
  Increase in the amplitude of the EMG response, with constant response latency, corresponding to the increase in the AMG response as stimulus strength (current) is increased.
Maximal EMG amplitude | During stimulation
  The observation of a maximal EMG amplitude, corresponding to the maximal AMG response, at maximal and supramaximal (up to maximal+10%, but below 70 mA) stimulus levels.
Consistency in amplitude | During stimulation
  Consistency in the amplitude of the AMG and EMG response amplitudes, with measured variations less than 10%, on repeated 1 Hz stimulation when the stimulus current is held constant between threshold and supramaximal intensity.
  Consistency of the AMG and EMG response amplitudes in repeated (ST and TOF) stimulus protocols (in which variation should be less than 10%).
  Consistency of EMG response characteristics and association with AMG responses independent of patient age, gender, or weight (despite different stimulus amplitudes being required to elicit submaximal and supramaximal responses).
  Consistency of EMG response characteristics and association with AMG responses independent of whether the right or left arm is being stimulated.
Discomfort level | During stimulation
  Establish the discomfort associated with nerve stimulation (from submaximal to supramaximal current amplitudes) in awake, unpremedicated human volunteers. Assessment will be made using an 11-point visual analog score (VAS) scale, anchored with 0 = no distress and 10 = worst distress ever experienced

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States